CLINICAL TRIAL: NCT02107716
Title: Will Adjusting the pH of Lidocaine Reduce the Pain During Injection of Local Anaesthetic?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 2013/2297A
Record Dates: First submitted 2014-04-04; First posted 2014-04-08 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Needlestick Injuries
Keywords: Pain; Injections; Lidocaine; Healthy volunteers
MeSH Terms: conditions — Needlestick Injuries; Pain | interventions — Lidocaine; Bicarbonates

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bicarbonate (Experimental): Each participant will receive two lidocaine injections on the abdomen with different pH
  Interventions: Procedure: Lidocaine injection with bicarbonate; Procedure: lidocaine injection

INTERVENTIONS:
Procedure: Lidocaine injection with bicarbonate — bicarbonate added to change pH
Procedure: lidocaine injection — Lidocaine injection with pH unchanged

SUMMARY:
This study will investigate the influence of adjusting the pH of lidocaine on pain during subcutaneous injection. Each participant will receive two injections on the abdomen with different pH. After each injection, the subject will be asked to evaluate the pain on a Visual analog scale (0-100 mm). It is anticipated that the pain decreases with increasing pH. The aim of the study is to find a simple method for pain reduction that can be used in clinical practice.

ELIGIBILITY:
Inclusion Criteria: fyll inn

* Age 18-65 years

Exclusion Criteria:

* Kidney, heart or liver disease
* Eczema or psoriasis on injection site
* Neuropathy
* Regular use of painkillers
* Hypersensitivity of Lidocaine
* Pregnancy
* Diabetes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-02; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Pain | 60 seconds
  1. Visual Analog Scale 0-100 mm
  2. Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Vilhjalmur Finsen, Prof md, Study Director — Norwegian University of Science and Technology
Locations (1):
- Department of Neuroscience, NTNU, Trondheim, Norway

REFERENCES:
- [Result] Skarsvag TI, Wago KJ, Tangen LF, Lundbom JS, Hjelseng T, Ballo S, Finsen V. Does adjusting the pH of lidocaine reduce pain during injection? J Plast Surg Hand Surg. 2015 Oct;49(5):265-267. doi: 10.3109/2000656X.2015.1047780. Epub 2015 May 19. PMID 25991379